CLINICAL TRIAL: NCT06146257
Title: A First-in-human, Phase 1, Dose Escalation and Expansion Study to Evaluate the Safety, Pharmacokinetics, Pharmacodynamics and Preliminary Efficacy of GLB-001 in Patients With Relapsed or Refractory Acute Myeloid Leukemia or Relapsed or Refractory Higher-risk Myelodysplastic Syndromes
Brief Title: A Study of GLB-001 in Patients With Relapsed or Refractory Acute Myeloid Leukemia or Relapsed or Refractory Higher Risk Myelodysplastic Syndromes
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: GluBio Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GLB-001-01
Record Dates: First submitted 2023-11-10; First posted 2023-11-24 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Acute Myeloid Leukemia; Myelodysplastic Syndromes
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dose Escalation of GLB-001 as a Monotherapy in Participants with R/R AML and R/R HR-MDS-Phase 1a (Experimental): Part 1a (Dose Escalation) of the study will enroll R/R AML and R/R HR-MDS participants and will evaluate the safety, tolerability, PK, PD and preliminary efficacy of GLB-001 administered orally, and determine the maximum tolerated dose/maximum administered dose (MTD/MAD) in R/R AML or R/R HR-MDS patients who are eligible for dose limiting toxicity (DLT) evaluation.
  Interventions: Drug: GLB-001
- Dose Expansion of GLB-001 as a Monotherapy in Participants with R/R AML and R/R HR-MDS-Phase 1b (Experimental): Part 1b (Dose Expansion) will confirm tolerability of the selected doses and schedules and evaluate whether efficacy is in a range that warrants further clinical development for R/R AML and R/R HR-MDS participants.
  Interventions: Drug: GLB-001

INTERVENTIONS:
Drug: GLB-001 — Administered orally according to the assigned treatment schedule
  Other Names: GLB-C183-A-2

SUMMARY:
Study GLB-001-01 is a first-in-human (FIH), Phase 1, open-label, dose escalation and expansion clinical study of GLB-001 in participants with relapsed or refractory acute myeloid leukemia (R/R AML) or in participants with relapsed or refractory higher-risk myelodysplastic syndromes (R/R HR-MDS). The dose escalation part (Phase 1a) of the study will evaluate the safety, tolerability, pharmacokinetics (PK), pharmacodynamics (PD) and preliminary efficacy of GLB-001 administered orally. Approximately 24 participants (up to 42 participants) may be enrolled in Phase 1a of the study.

The dose expansion part (Phase 1b) will be followed to understand the relationships among dose, exposure, toxicity, tolerability and clinical activity, to identify minimally active dose, and to select the recommended dose(s) for phase 2 study. Up to 24 participants (12 participants per dose level) may be enrolled in Phase 1b of the study.

DETAILED DESCRIPTION:
A standard 3+3 dose-escalation design will be applied to evaluate a set of several dose levels to determine the maximum tolerated dose (MTD) or maximum administered dose (MAD) of GLB-001 in R/R AML or R/R HR-MDS patients who are eligible for DLT evaluation. The actual dose-escalation magnitude or dosing frequency may be adjusted based on the available PK and safety data in human.

After the MTD or MAD of GLB-001 is defined in Phase 1a, 1 or 2 dose levels will be selected for expansion per safety review committee (SRC) recommendation, approximately 12 patients will be enrolled per dose level. Recommended phase 2 dose (RP2D) will be selected based on the results of PK, PD, safety and efficacy in the dose escalation and expansion study.

ELIGIBILITY:
Inclusion Criteria:

* Participants is ≥ 18 years of age at the time of signing the Informed Consent Form (ICF).
* Participants must understand and voluntarily sign an ICF prior to any study-related assessments/procedures being conducted.
* Participants are willing and able to adhere to the study visit schedule and other protocol requirements.
* Participants with histologically or cytologically confirmed AML including de novo AML or secondary AML transformed from MDS according to 2022 World Health Organization (WHO) criteria classification, or with histologically or cytologically confirmed HR-MDS.
* R/R AML and R/R HR-MDS who have failed or are ineligible for all available therapies which may provide clinical benefit.
* Participants must have the following screening laboratory values:

  * Total white blood cell count (WBC) < 25 x 10^9/L prior to the first dose of the study drug.
  * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 3.0 × upper limit of normal (ULN), unless considered due to extensive leukemic liver involvement, in which case AST and ALT can be ≤ 5.0 x ULN.
  * Serum total bilirubin ≤ 1.5 x ULN, unless considered due to Gilbert's syndrome, in which case serum total bilirubin < 3 x ULN.
  * Estimated serum creatinine clearance of ≥ 60 mL/min using the Cockcroft-Gault equation. Measured creatinine clearance from a 24-hour urine collection is acceptable if clinically indicated.
  * International normalized ratio (INR) ≤ 1.5 x ULN and active partial thromboplastin time (aPTT) ≤ 1.5 x ULN.
* Life expectancy ≥ 12 weeks.
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 to 2.
* Female Participants of child-bearing potential must have a negative serum or urine pregnancy test at screening and at pre-dose on Cycle 1 Day 1 (C1D1).

Exclusion Criteria:

* Participants with acute promyelocytic leukemia (APML).
* Participants with known leukemic involvement in central nervous system (CNS).
* Receipt of anticancer medications/therapies within 5 half-lives or 28 days before the first administration of the study drug.
* Participants with unresolved clinically significant non-hematologic toxicities of ≥ Grade 2 AE from prior therapies with exception of residual alopecia.
* Participants with chronic graft versus host disease (GVHD) requiring systemic immunosuppressive therapy.
* Participants with active malignancies other than AML or MDS.
* Participants who have undergone major surgery ≤ 4 weeks prior to the first dose of the study drug.
* Participants with immediately life-threatening, severe complications of leukemia such as disseminated/uncontrolled infection (bacterial and/or fungal), uncontrolled bleeding, and/or uncontrolled disseminated intravascular coagulation.
* Participants with known chronic, active infection of hepatitis B virus (HBV), hepatitis C virus C (HCV), human immunodeficiency virus (HIV).
* Participants unable to swallow oral medications, or Participants with clinically significant diarrhea, vomiting or malabsorption felt limited absorption of orally administered medications.
* Participants with any other significant medical conditions, any other conditions, laboratory abnormality, or psychiatric illness which place the Participants at unacceptable risk if he/she were to participate in the study or that would hamper the Participants understanding of the study, or would prevent the Participant from complying with the study.
* Medications or supplements that are known to be strong and moderate inhibitors or inducers of CYP450 isozyme 3A4 (CYP3A4) and/or P-glycoprotein (P-gp), or strong inhibitors or inducers of CYP450 isozyme 2C8 (CYP2C8) within 14 days or 5 half-lives, whichever is shorter, before the first dose of study drug.
* Pregnant or lactating women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2024-01-11 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-10-08 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting Toxicity (DLT) | Up to 28 days after first dose of study treatment in Phase 1a
  Dose-limiting toxicity is defined as the treatment emergent adverse events (TEAEs) meeting protocol specified DLT criteria and occurring within the DLT assessment period.
Maximum Tolerated Dose (MTD)/Maximum Administered Dose (MAD) | Up to 2 years
  Maximum tolerated dose is defined as the highest dose level at which no more than 1 of 6 DLT-evaluable participants experienced a DLT. If MTD is not established at the end of dose escalation phase, the maximum safety dose will be defined as Maximum administered dose.
Incidence of Adverse Events (AEs) | Up to 2 years
  Adverse Events will be graded according to the National Cancer Institute Common Terminology Criteria for AE (NCI CTCAE) version 5.0.
Recommended Phase 2 Dose (RP2D) | Up to 2 years
  Recommended phase 2 dose based on the totality of data across dosing cohorts in the dose escalation and expansion phases of the study including PK, PD, safety and efficacy outcomes.

SECONDARY OUTCOMES:
GLB-001 Pharmacokinetics-AUC0-last | Up to 2 years
  Area under the concentration-time curve from zero to the last measurable concentration.
GLB-001 Pharmacokinetics-AUC0-24 | Up to 2 years
  Area under the concentration-time curve from 0 to 24 hours.
GLB-001 Pharmacokinetics-AUC0-∞ | Up to 2 years
  Area under the concentration-time curve from 0 to infinity.
GLB-001 Pharmacokinetics-Cmax | Up to 2 years
  Maximum plasma concentration.
GLB-001 Pharmacokinetics-Tmax | Up to 2 years
  The time to reach maximum concentration.
GLB-001 Pharmacokinetics-T1/2 | Up to 2 years
  Terminal half-life.
GLB-001 Pharmacokinetics-Vd/F | Up to 2 years
  Apparent volume of distribution.
GLB-001 Pharmacokinetics-LI | Up to 2 years
  Linear index.
GLB-001 Pharmacokinetics-CL/F | Up to 2 years
  Apparent clearance.
GLB-C183-A-2R (Isomer of GLB-001) Pharmacokinetics-AUC0-last | Up to 2 years
  Area under the concentration-time curve from zero to the last measurable concentration.
GLB-C183-A-2R Pharmacokinetics-AUC0-24 | Up to 2 years
  Area under the concentration-time curve from 0 to 24 hours.
GLB-C183-A-2R Pharmacokinetics-AUC0-∞ | Up to 2 years
  Area under the concentration-time curve from 0 to infinity.
GLB-C183-A-2R Pharmacokinetics-Cmax | Up to 2 years
  Maximum plasma concentration.
GLB-C183-A-2R Pharmacokinetics-Tmax | Up to 2 years
  The time to reach maximum concentration.
GLB-C183-A-2R Pharmacokinetics-T1/2 | Up to 2 years
  Terminal half-life.
GLB-C183-A-2R Pharmacokinetics-Vd/F | Up to 2 years
  Apparent volume of distribution.
GLB-C183-A-2R Pharmacokinetics-LI | Up to 2 years
  Linear index.
GLB-C183-A-2R Pharmacokinetics-CL/F | Up to 2 years
  Apparent clearance.
Complete Remission Without Minimal Residual Disease (CRMRD-) Rate in Participants with Acute Myeloid Leukemia (AML) | Up to 2 years
  CRMRD- rate is defined as the percent of participants with minimal residual disease negative complete remission. CRMRD- will be assessed by the 2022 European Leukemia Net Response Criteria (2022 ELN) for AML .
Complete Remission (CR) Rate in Participants with AML | Up to 2 years
  CR rate is defined as the percent of participants whose best response is CR. CR will be assessed by 2022 ELN for AML.
CR with Incomplete Hematologic Recovery (CRi) Rate in Participants with AML | Up to 2 years
  CRi rate is defined as the percent of participants whose best response is CRi. CRi will be assessed by 2022 ELN for AML.
CR with Partial Hematological Recovery (CRh) Rate in Participants with AML | Up to 2 years
  CRh rate is defined as the percent of participants whose best response is CRh. CRh will be assessed by 2022 ELN for AML.
Morphologic Leukemia-free State (MLFS) Rate in Participants with AML | Up to 2 years
  MLFS rate is defined as the percent of participants with the best response of morphologic leukemia-free state. MLFS will be assessed by 2022 ELN for AML.
Partial Remission (PR) Rate in Participants with AML | Up to 2 years
  PR rate is defined as the percent of participants whose best response is PR. PR will be assessed by 2022 ELN for AML.
Duration of Remission or Response (DOR) in Participants with AML | Up to 2 years
  For participants with best response of any of CRMRD-, CR, CRh, CRi, PR, and MLFS, DOR is measured from the time when criteria (2022 ELN for AML) for the best response of any of CRMRD-, CR, CRh, CRi, PR, and MLFS are first met (whichever is first recorded) until the first date at which relapse, or progressive disease is objectively documented assessment.
Time to Remission or Response (TOR) in Participants with AML | Up to 2 years
  Time to onset of first remission or response is defined as the time interval from the date of first dose and the earliest date any remission or response [any CRs (including CR, CRh and CRi) or PR] is observed.
Stable Disease (SD) Rate in Participants with AML | Up to 2 years
  SD rate is defined as the percent of participants with the best response of stable disease. SD will be assessed by 2022 ELN for AML.
CR Rate in Participants with Higher Risk Myelodysplastic Syndromes (HR-MDS) | Up to 2 years
  CR rate is defined as the percent of participants whose best response is CR. CR will be assessed by 2006 Modified International Working Group (IWG) MDS response criteria.
PR Rate in Participants with HR-MDS | Up to 2 years
  PR rate is defined as the percent of participants whose best response is PR. PR will be assessed by 2006 Modified IWG MDS response criteria.
SD Rate in Participants with HR-MDS | Up to 2 years
  SD rate is defined as the percent of participants with the best response of stable disease. SD will be assessed by 2006 Modified IWG MDS response criteria.
DOR in Participants with HR-MDS | Up to 2 years
  For participants with best response of any of CR, marrow CR, or PR, DOR is measured from the time when criteria (2006 Modified IWG MDS response criteria) for the best response of any of CR, marrow CR, or PR are first met (whichever is first recorded) until the first date at which relapse or progressive disease is objectively documented assessment.
TOR in Participants with HR-MDS | Up to 2 years
  Time to onset of first remission or response is defined as the time interval from the date of first dose of GLB-001 and the earliest date any remission or response [any CRs (including CR, marrow CR or PR)] is observed.
Progression-free Survival (PFS) in Participants with AML or HR-MDS | Up to 2 years
  PFS is defined as the time from the first dose of GLB-001 to the first occurrence of relapse or progression or death from any cause.
Overall Survival (OS) in Participants with AML or HR-MDS | Up to 2 years
  OS is defined as the time from the first dose of GLB-001 to death due to any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Gang Lu, Ph.D., Study Director — GluBio Therapeutics Inc.
Locations (8):
- United States (8):
  - City of Hope Medical Center, Duarte, California
  - University of California Irvine, Irvine, California
  - University of Kansas Medical Center Research Institute, Inc., Kansas City, Kansas
  - Alliance for Multispecialty Research, LLC, Merriam, Kansas
  - Roswell Park Comprehensive Cancer Center, Buffalo, New York
  - Memorial Sloan Kettering Cancer Center-David H. Koch Center, New York, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - University of Texas M. D. Anderson Cancer Center, Houston, Texas